CLINICAL TRIAL: NCT01207765
Title: A Phase II, Safety and Efficacy Study of Fixed Dose Radioimmunotherapy (Zevalin, Yttrium-90 Ibritumomab Tiuxetan) for Patients With Incomplete Response to Chemotherapy Prior to Autologous Stem Cell Transplant for Multiple Myeloma
Brief Title: Zevalin for Patients With Incomplete Response to Chemo Prior to Autologous Stem Cell Transplant for Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: changes in practice
Sponsor: Tufts Medical Center (Other)
Collaborators: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zevalin
Record Dates: First submitted 2010-09-21; First posted 2010-09-23 (Estimated); Results first posted 2016-10-28 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-02

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Zevalin
MeSH Terms: conditions — Multiple Myeloma | interventions — ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zevalin (Experimental): 1.5mg of 111In Zevalin (containing 5 mCi of 111In) will be used for radioimaging on study day +1. 90Y Zevalin will be administered seven to nine days after 111In Zevalin administration. The dose of 90Y Zevalin will be 0.4 mCi/kg, capped at a maximum dose of 32 mCi.
  Interventions: Drug: indium-111-ibritumomab tiuxetan; Drug: 90Y Zevalin

INTERVENTIONS:
Drug: indium-111-ibritumomab tiuxetan — 1.5mg of 111In Zevalin (containing 5 mCi of 111In) will be used for radioimaging. 111In Zevalin will be administered by a 10 minute slow IV push injection immediately following completion of the rituximab infusion. 111In Zevalin may be injected by stopping the flow from the IV bag and injecting the radiolabeled antibody directly into the IV line. A 0.22 micron filter must be on line between the drug infusion port and the patient. The line must be flushed with at least 10cc of normal saline after 111In Zevalin has been injected.
  Other Names: 111 In Zevalin
Drug: 90Y Zevalin — Each patient will receive a single therapeutic dose of 90Y Zevalin at a dose of 0.4 mCi/kg, capped at a maximum dose of 32 mCi. 90Y Zevalin will be administered intravenously as a slow IV push over 10 minutes. 90Y Zevalin may be directly infused by stopping the flow from the IV bag and injecting the radiolabeled antibody directly into the IV line. A 0.22 micron filter must be on line between the syringe and the infusion port. The line must be flushed with at least 10cc normal saline after 90Y Zevalin has been infused.

SUMMARY:
The study involves the use of a targeted form of radiation, in addition to standard high dose chemotherapy and stem cell transplant for multiple myeloma. The use of targeted radiation is designed to kill more multiple myeloma cells while avoiding the side effects of standard radiation. This type of targeted radiation (also known as radioimmunotherapy) has been approved by the Food and Drug Administration (FDA) for the treatment of a related disease, lymphoma under the trade name, Zevalin©. Zevalin© has been added to high dose chemotherapy and stem cell transplants for patients with lymphoma and is now being studied in this clinical trial for patients with multiple myeloma. This trial is only available at Tufts Medical Center.

The proposed clinical trial will test whether CD20-targeted radio-immunotherapy can be safe and effective when integrated into a standard regimen of myeloablative chemotherapy and autologous stem cell rescue in patients with measurable disease prior to high dose chemotherapy and autologous stem cell transplant for multiple myeloma.

DETAILED DESCRIPTION:
Patients with multiple myeloma scheduled for standard of care high dose melphalan and autologous stem cell transplant who have an incomplete response to induction treatment (i.e. with measurable disease) following peripheral blood stem cell collection are candidates for participation on this trial. 90Y Zevalin targets CD20 expressed on the surface of mature B-cells and is FDA approved for relapsed/refractory low grade lymphoma. This is a single arm, phase II safety and efficacy study of 90-Y Zevalin in multiple myeloma. Subjects will receive cold antibody (Rituximab 100mg/m2) followed by 5 mCi test dose of 111-In Zevalin on transplant day -21. Gamma camera images are obtained 48 to 72 hours after 111-In Zevalin to document appropriate / expected distribution of radiotracer. On transplant day -14, subjects will receive another cold antibody dose followed by 90Y Zevalin 0.4 mg/kg (max 32 mCi) as single dose. Subjects are admitted for transplant on day -3 and proceed with institution standard high dose melphalan (200mg/m2) on day -2. Subjects are followed for safety for 6 weeks after transplant.

ELIGIBILITY:
Inclusion Criteria:

* Meet established criteria for the diagnosis of multiple myeloma
* Durie-Salmon stage II or III disease
* Measurable disease in the serum and/or urine
* Scheduled to receive high dose chemotherapy and autologous stem cell transplant for multiple myeloma
* Individuals who have previously undergone autologous stem cell transplant are eligible for this study provided more than 6 months have elapsed from the prior transplant.
* Minimum stem cell dose of 4x106 CD34+ MNC / kg stored for autologous stem cell rescue.
* Adequate hematologic reserve as evidenced by ANC ≥ 1500/mm3 and platelets ≥ 100,000/mm3.
* Serum direct bilirubin ≤ 2.0 mg/dl and transaminases ≤ 3x institution upper limit of normal.
* Serum creatinine ≤ 2 mg/dl with creatinine clearance ≥ 60 ml/min (either calculated or measured).

Exclusion Criteria:

* Stage I or smoldering myeloma, isolated plasmacytoma, or benign monoclonal gammopathy
* Non-secretory multiple myeloma
* Pregnant or lactating women
* Males and females who do not agree to practice approved methods of birth control for the duration of the study
* Presence of active infection
* Receipt of previous radiation therapy to critical organs exceeding any of the following limits: kidney 500 cGy, liver 1000 cGy, lungs 500 cGy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-04; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas K Klein, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Attal M, Harousseau JL, Stoppa AM, Sotto JJ, Fuzibet JG, Rossi JF, Casassus P, Maisonneuve H, Facon T, Ifrah N, Payen C, Bataille R. A prospective, randomized trial of autologous bone marrow transplantation and chemotherapy in multiple myeloma. Intergroupe Francais du Myelome. N Engl J Med. 1996 Jul 11;335(2):91-7. doi: 10.1056/NEJM199607113350204. PMID 8649495
- [Background] Moreau P, Facon T, Attal M, Hulin C, Michallet M, Maloisel F, Sotto JJ, Guilhot F, Marit G, Doyen C, Jaubert J, Fuzibet JG, Francois S, Benboubker L, Monconduit M, Voillat L, Macro M, Berthou C, Dorvaux V, Pignon B, Rio B, Matthes T, Casassus P, Caillot D, Najman N, Grosbois B, Bataille R, Harousseau JL; Intergroupe Francophone du Myelome. Comparison of 200 mg/m(2) melphalan and 8 Gy total body irradiation plus 140 mg/m(2) melphalan as conditioning regimens for peripheral blood stem cell transplantation in patients with newly diagnosed multiple myeloma: final analysis of the Intergroupe Francophone du Myelome 9502 randomized trial. Blood. 2002 Feb 1;99(3):731-5. doi: 10.1182/blood.v99.3.731. PMID 11806971
- [Background] Treon SP, Pilarski LM, Belch AR, Kelliher A, Preffer FI, Shima Y, Mitsiades CS, Mitsiades NS, Szczepek AJ, Ellman L, Harmon D, Grossbard ML, Anderson KC. CD20-directed serotherapy in patients with multiple myeloma: biologic considerations and therapeutic applications. J Immunother. 2002 Jan-Feb;25(1):72-81. doi: 10.1097/00002371-200201000-00008. PMID 11924912
- [Background] Matsui W, Wang Q, Barber JP, Brennan S, Smith BD, Borrello I, McNiece I, Lin L, Ambinder RF, Peacock C, Watkins DN, Huff CA, Jones RJ. Clonogenic multiple myeloma progenitors, stem cell properties, and drug resistance. Cancer Res. 2008 Jan 1;68(1):190-7. doi: 10.1158/0008-5472.CAN-07-3096. PMID 18172311
- [Background] Blade J, Samson D, Reece D, Apperley J, Bjorkstrand B, Gahrton G, Gertz M, Giralt S, Jagannath S, Vesole D. Criteria for evaluating disease response and progression in patients with multiple myeloma treated by high-dose therapy and haemopoietic stem cell transplantation. Myeloma Subcommittee of the EBMT. European Group for Blood and Marrow Transplant. Br J Haematol. 1998 Sep;102(5):1115-23. doi: 10.1046/j.1365-2141.1998.00930.x. No abstract available. PMID 9753033
- [Background] Knox SJ, Goris ML, Trisler K, Negrin R, Davis T, Liles TM, Grillo-Lopez A, Chinn P, Varns C, Ning SC, Fowler S, Deb N, Becker M, Marquez C, Levy R. Yttrium-90-labeled anti-CD20 monoclonal antibody therapy of recurrent B-cell lymphoma. Clin Cancer Res. 1996 Mar;2(3):457-70. PMID 9816191

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zevalin
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Simon two-stage, min-max design test the hypothesis H0: p</=0.05 (the expected response rate for no treatment) versus Ha: p>/=0.30 (a clinically significant response rate) with a=0.05 and b=0.20.
Arm/Group | Zevalin
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Safety and Efficacy
Description: Efficacy: objective response rate (CR + PR) at 12 and 104 days following radioimmunotherapy. Safety: the rate of occurrence of defined toxic events including non-engraftment and unacceptable biodistribution of 90Y Zevalin occurring by day +42 following transplant. Response determined according to Blade' Criteria (Bladé J, Br J Haematol.1998 Sep;102(5):1115-23) for multiple myeloma; Response based on reduction of monoclonal protein (M-protein) from initial presentation.
Time Frame: Through day +104 following immunotherapy
Population: 6 subjects had objectively measurable disease and were evaluable for response, 8 subjects received study intervention and are evaluable for safety
Measure: Number; unit: participants
Groups:
- Zevalin: 90Y Zevalin: Each patient will receive a single therapeutic dose of 90Y Zevalin at a dose of 0.4 mCi/kg, capped at a maximum dose of 32 mCi.
Arm/Group | Zevalin
Number analyzed (Participants) | 8
participants
  CR/PR at +12 days: number analyzed (Participants) | 6
  CR/PR at +12 days | 1
  CR/PR at +104 days: number analyzed (Participants) | 6
  CR/PR at +104 days | 5
  Participants with toxic events | 5

2. Secondary Outcome: Time to Engraftment in Patients Who Proceed to Myeloablative Chemotherapy After Receiving 90Y Zevalin® (Ibritumomab Tiuxetan).
Description: Number of days from stem cell infusion (day +0) to day of neutrophil engraftment (first of three consecutive days with absolute neutrophil count > 500)
Time Frame: Transplant through day 42
Population: Analyzed on intent-to-treat basis
Measure: Median (Full Range); unit: Days
Arm/Group | Zevalin
Number analyzed (Participants) | 8
Days | 13 [9 to 31]

3. Secondary Outcome: Degree of CD20 Expression on Plasma Cells and/or Targeting of Post-germinal Center B Cells Correlation With Toxicity, Response and Biodistribution
Description: CD20 immunohistochemical staining of plasma cells on baseline bone marrow biopsy specimen, graded on qualitative scale (0 to +++)
Time Frame: 2 weeks prior - 2 weeks post transplant
Population: Immunohistochemical analysis showed inconsistent / insufficient CD20 staining on surface of plasma cells; comparisons could not be made
Arm/Group | Zevalin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Zevalin
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zevalin (N=8)
Septic thrombophlebitis (Blood and lymphatic system disorders) | 1 (1)
Perianal absess (Infections and infestations) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zevalin (N=8)
MRSA bacteremia (Infections and infestations) | 1 (1)
S. viridans bacteremia (Infections and infestations) | 1 (1)
S. epidermitis (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Study ended at end of stage 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes